CLINICAL TRIAL: NCT05328284
Title: PASTE: PASCAL for Tricuspid Regurgitation - a European Registry
Brief Title: PASCAL for Tricuspid Regurgitation - a European Registry
Acronym: PASTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Jörg Hausleiter, Deputy chief, LMU Klinikum
Other Study IDs: 21-0385
Record Dates: First submitted 2022-03-15; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PASCAL: patients treated with PASCAL leaflet repair system in the treatment of TR in a commercial use setting
  Interventions: Device: PASCAL leaflet repair system

INTERVENTIONS:
Device: PASCAL leaflet repair system — transcatheter Implantation of one or more PASCAL devices in the tricuspid valve

SUMMARY:
This study aims to investigate the safety and efficacy of the PASCAL leaflet repair system in the treatment of tricuspid regurgitation in a commercial use setting including all consecutive patients at the participating Centers in an observational fashion.

DETAILED DESCRIPTION:
Tricuspid regurgitation (TR) is associated with high morbidity and mortality, but many patients are ineligible for surgical treatment due to age and co-morbidities. As a consequence, transcatheter treatment techniques have evolved over the last years. Leaflet repair is one of the most commonly used techniques and has recently gained commercial approval for dedicated TR treatment. The PASCAL (Edwards Lifesciences, Irvine, USA) offers the possibility for independent leaflet grasping and a central spacer can bridge larger coaptation gaps. The hitherto evidence is mainly based on compassionate use data. This study aims to report the first commercial use in a multicenter study with a large patient cohort und long-term follow-up.

Aim of the study is to investigate safety and efficacy of the PASCAL leaflet repair system in the treatment of TR in a commercial use setting.

Study design is a multicenter, single-device, retro- and prospective, observational registry. All consecutive patients undergoing treatment with the PASCAL system for tricuspid regurgitation in a commercial setting are included.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with the PASCAL system for tricuspid regurgitation in a commercial setting

Exclusion Criteria:

* Patient age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients that have undergone transcatheter tricuspid valve repair with the PASCAL system since its commercial approval in 02/2019 at the participating centres shall be included in the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Change of TR severity | 1 year
  TR ≤ grade 2+ (moderate)

SECONDARY OUTCOMES:
Rate of technical success | 1 day
  absence of procedural mortality, successful access, delivery and retrieval of the delivery system, successful deployment and positioning, freedom from emergency surgery
Rate of procedural safety | 1 week
  Absence of periprocedural and in-hospital adverse events
New York Heart Association (NYHA) functional class | 1 year
  Level of exertional dyspnea (I - IV)
6-minute walk distance (6MWD) | 1 year
  physical capacity measured by 6MWD in meters
NT-proBNP level | last available follow-up (at least 1 year after intervention)
  cardiac biomarker level (in pg/nl)
right heart dimension | 1 year
  Right ventricular end-diastolic Diameter (in mm)
right heart function | 1 year
  tricuspid annular plane systolic excursion (TAPSE, in mm)
tricuspid regurgitation severity | last available follow-up (at least 1 year after intervention)
  TR severity grading on a five-grade scheme (1-5)
transtricuspid gradient | 1 year
  transvalvular antegrade gradient over tricuspid valve (in mmHg)
pulmonary artery pressure (PAP) | 1 year
  estimated PAP by echocardiography (in mmHg)
inferior vena cava (IVC) dimension | 1 year
  IVC Diameter during expiration (in mm)

CONTACTS AND LOCATIONS:
Locations (14):
- Germany (11):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herz & Diabeteszentrum Nordrhein Westfalen, Bad Oeynhausen
  - Universitätsklinikum Essen, Essen
  - Marienkrankenhaus Hamburg, Hamburg
  - Universitäres Herz- und Gefäßzentrum Hamburg, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Herzzentrum Leipzig, Leipzig
  - LMU University Hospital, Munich
  - Universitätsklinikum Siegburg, Siegburg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinik Ulm, Ulm
- Karolinska University Hospital, Stockholm, Sweden
- Switzerland (2):
  - Inselspital Bern, Bern
  - Kantonsspital Luzern LUKS, Lucerne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wild MG, Stolz L, Rosch S, Rudolph F, Goebel B, Koll B, von Stein P, Rottbauer W, Rassaf T, Beucher H, Kraus M, Kassar M, Geisler T, Ruck A, Ferreira-Martins J, Toggweiler S, Sagmeister P, Westermann D, Stocker TJ, Weckbach LT, Nabauer M, Settergren M, Dawkins S, Kister T, Praz F, Vorpahl M, Konstandin MH, Ludike P, Kessler M, Iliadis C, Kalbacher D, Lauten P, Gercek M, Besler C, Lurz P, Hausleiter J; PASTE Investigators. Transcatheter Valve Repair for Tricuspid Regurgitation: 1-Year Results From a Large European Real-World Registry. J Am Coll Cardiol. 2025 Jan 28;85(3):220-231. doi: 10.1016/j.jacc.2024.10.068. Epub 2024 Oct 28. PMID 39466215